CLINICAL TRIAL: NCT00063037
Title: Building Better Bones in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: R01HD037748 (NIH)
Record Dates: First submitted 2003-06-19; First posted 2003-06-20 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-05

CONDITIONS: Osteoporosis
Keywords: Bone mass; Calcium intake; Prevention of osteoporosis; Optimizing peak bone mass; Bone mineral density
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Behavioral: Behavioral modification - nutrition education

SUMMARY:
Calcium is important for healthy bone growth in children. Poor bone growth and development during childhood can lead to osteoporosis later in life. This study will evaluate a nutrition education program designed to increase the amount of calcium children receive. The study will determine whether the program will result in long-term dietary changes and healthier bones in children.

DETAILED DESCRIPTION:
Increased calcium intake is effective in increasing bone mineral density in children, but the effect disappears when calcium supplements are discontinued. Increased dietary calcium from daily food sources may have a greater impact on bone density than that achieved by calcium supplements. However, studies have not yet demonstrated sustained achievement of increased calcium from food sources. In addition, the effects of baseline calcium intake, bone density, and puberty status may influence bone response to increased dietary calcium. This study will develop, implement, and evaluate a Behavioral Modification-Nutrition Education (BM-NE) Intervention Program designed to promote sustained increases in dietary calcium. The study will quantify the impact of increased dietary calcium on bone density during growth and development and will determine whether the presence of risk factors for low bone density influences compliance with the program.

Participants will be recruited into two groups: a group of healthy children with no known risk factors for low bone density (i.e., no known chronic disease or previous oral steroid exposure), and a group of healthy children with potential risk factors for low bone density (previous fracture from usual childhood activities, daily dietary calcium refusal, lactose intolerance, family history of osteoporosis). Children with and without risk factors will be randomly assigned to participate in an intensive BM-NE intervention group or a usual care group that will receive counseling on bone health. The BM-NE Program will consist of five group sessions for parents and children over 6 weeks. The program will use individualized plans to increase children's calcium intake to 1500 mg per day.

Children will be followed for 3 years. Primary outcome measures will include daily calcium intake and bone mineral density. Data on height, weight, sexual and skeletal maturation, and physical activity will also be collected.

ELIGIBILITY:
Inclusion Criteria

* Height or weight above the third percentile for age
* Normal weight (< 130% of desirable body weight)
* English speaking

Exclusion Criteria

* Significant health condition
* Medication known to affect growth (e.g., thyroxin, growth hormone, steroid medication)
* Ritalin or Adderall medication
* Significant developmental or delay impairment (e.g., autism, cerebral palsy, mental retardation)

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 139
Dates: Start 1999-06; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Babette Zemel, Ph.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Weber DR, Stark LJ, Ittenbach RF, Stallings VA, Zemel BS. Building better bones in childhood: a randomized controlled study to test the efficacy of a dietary intervention program to increase calcium intake. Eur J Clin Nutr. 2017 Jun;71(6):788-794. doi: 10.1038/ejcn.2017.5. Epub 2017 Feb 22. PMID 28225052